CLINICAL TRIAL: NCT04234230
Title: Improved Health Care for People With Chronic Heart Disease and Implanted Cardiac Support Through Curricular Self-management - Phase 1: Prevalence Study
Brief Title: Improved Self-management for Patients on Ventricular Assist Device (VAD)
Acronym: SELMA
Status: Completed | Type: Observational
Sponsor: University of Freiburg (Other)
Collaborators: University Heart Center Freiburg - Bad Krozingen (Other); Heart and Diabetes Center North-Rhine Westfalia (Other); German Heart Center (Other); Heart Center Leipzig - University Hospital (Other)
Responsible Party: Principal Investigator, Christiane Kugler, Professor Doctor. rer. biol. hum., University of Freiburg
Other Study IDs: 01VSF18012
Record Dates: First submitted 2019-10-02; First posted 2020-01-21 (Actual); Last update posted 2020-11-06 (Actual); Status verified 2020-11

CONDITIONS: Ventricular Assist Device; Self-management; Psychological Factors
Keywords: Ventricular Assist Device; Self-management; Psychosocial Factors
MeSH Terms: interventions — Contraceptive Prevalence Surveys

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- VAD Patients: Patients with implanted ventricular assist device in the outpatient setting
  Interventions: Other: Prevalence Survey

INTERVENTIONS:
Other: Prevalence Survey — Questionnaire survey on self-management

SUMMARY:
The number of patients with end-stage heart disease requiring the implantation of ventricular assist devices (VAD) is steadily increasing. Living with a VAD exposes the patients to multiple challenges and the need to learn complex self-management skills. Inadequate self-management can lead to serious complications (e.g. bleeding or wound infections) and impair the psychosocial outcome. This study aims to provide multi-centered actual analysis of self-management capabilities as well as analyzing moderating predictors in VAD patients through standardized prevalence assessment. Using a cross-sectional design, this prevalence study will be conducted at four established German heartcenters (Freiburg, Berlin, Bad Oeynhausen, Leipzig). VAD-patients are questioned about their self-management skills using standardized Patient-reported outcome (PRO) measures. Secondary PRO measures include health-related quality of life, symptoms of anxiety and depression, post-traumatic stress symptoms, social support, and changed body-image. Relevant complications (bleeding, wound infections, thromboembolic neurological events) are taken from the patient records. Based on a conservative sample size estimation inclusion of 450 patients is envisioned. The expected results may contribute to an improved assessment of the current situation in terms of self-management skills and needs for curricular training concepts and psychosocial concomitant therapy. Long-term, the study results contribute to improve the health care for long-term VAD patients.

DETAILED DESCRIPTION:
The number of patients with end-stage heart disease requiring the implantation of ventricular assist devices (VAD) is steadily increasing. Due to advanced compensatory technological developments, VAD support has been established as a recognized therapy concept for the long-term care of those affected. Indications include a multi-year bridging therapy (up to 10 years) and increasingly a destination therapy. The Euromacs Register published the second report in 2018 and reported 2,947 registered VAD implantations in 2016 (+257 percent). Euromacs further points to a rising trend and demand for the use of VAD systems. In Germany, an increase of VAD implantation by 36.6 percent has been reported since 2011. The position paper of the German Society of Cardiology (2016) points to the fact that the range of indications for VAD implantation for patients with chronic heart disease will continue to change. The ISHLT Guideline (International Society for Heart and Lung Transplantation), published in 2018, calls for psychosocial care and standardized self-management skills for patients before, during, and in the long-term after VAD implantation. This is currently being implemented inconsistently in terms of structure and quality in German cardiac centers. After VAD implantation, patients and their relatives must be able to follow a complex therapeutic regimen. They need comprehensive knowledge as well as self-management skills for the safe management of everyday life in a domestic setting. These self-management capabilities include the so-called device handling (for example dealing with the technical equipment including battery replacement and controller monitoring), to perform the wound care of the driveline, to carry out anticoagulation measurements and adapted revenues of oral anticoagulant, to take further medication, to monitor vital signs (for example blood pressure, temperature) and, in the case of symptoms, to take adequate measures to prevent further complications (for example prompt information from the heart center on the onset of symptoms). In addition, lifestyle changes are an essential part of the success of long-term therapy. This requires a sufficient degree of self-management ability and mental stability. In addition, it is important to emotionally accept the dependence of a device on the heart, the changed body image, to cope with fears of (real potential) malfunctions and complications and to build up a subjective quality of life with a constant, visible and tangible companion at heart. The mental health of all those affected is considered to be in need of observation, although there is currently no reliable prevalence data on mental disorders. In a first survey in 2006, 64% had at least one psychologically / psychiatric treatment requiring diagnosis. All this shows, the challenges VAD patients have to face are complex. Thus, this study aims to provide multi-centered actual analysis of self-management capabilities as well as analyzing moderating predictors in VAD patients through standardized PRO prevalence assessment. The prevalence survey should be conducted in all outpatients (at least 3 months up to a maximum of 3 years at the VAD) in four established German cardiac centers (Freiburg, Berlin, Bad Oeynhausen, Leipzig). The study focuses on those involved in outpatient care, as they had to integrate the VAD into their daily lives after implantation and are able to report deficits, resources and needs on the basis of their experience of self-management. As an assessment instrument a standardized PRO measure was chosen to identify self-management skills and needs. Secondary PRO measures include health-related quality of life, symptoms of anxiety, depression and post-traumatic stress, as well as social support. Relevant complications (bleeding, wound infections, thromboembolic neurological events) are taken from the patient records. Based on a conservative sample size estimation inclusion of 450 patients is envisioned. The expected results may contribute to an improved assessment of the current situation in terms of self-management skills and needs for curricular training concepts and psychosocial concomitant therapy. Long-term, the study results contribute to improve the health care for long-term VAD patients. The study is planned to continue in a second and third phase to develop and test a standardized self-management care for VAD patients in Germany.

ELIGIBILITY:
Inclusion Criteria:

* Outpatient at the respective heart center
* Living in a home environment
* On device between 3 months and 3 years
* 18 years and older
* No contraindications (e.g. cognitive, language)
* Signed Informed Consent

Exclusion Criteria:

* In-patient stay
* Not living in a home environment (e.g. assisted living)
* On device less than 3 months or more than 3 years
* Underage
* Contraindications (e.g. cognitive, language)
* No signed Informed Consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients implanted with a ventricular assist device in the outpatient setting of four heart centers in Germany (Freiburg, Berlin, Bad Oeynhausen and Leipzig).
Sampling Method: Non-Probability Sample
Enrollment: 393 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2020-08-31 (Actual); Study Completion 2020-09-30 (Actual)

PRIMARY OUTCOMES:
Self-management Skills | October 2019 till January 2020
  As an assessment instrument a standardized PRO measure was chosen to identify self-management skills and needs.

SECONDARY OUTCOMES:
Health-related Quality of Life | October 2019 till January 2020
  The experienced health-related quality of life of the participants measured with a selfassessment questionnaire (QoL-VAD, KCCQ).
Social Support | October 2019 till January 2020
  The experienced social support of the participants measured with a selfassessment questionnaire (F-SozU).
Symptoms of Anxiety | October 2019 till January 2020
  Symptoms of anxiety measured via screening tool (HADS).
Symptoms of Depression | October 2019 till January 2020
  Symptoms of depression measured via screening tool (HADS, PHQ-9).
Symptoms of Posttraumatic Stress Disorder | October 2019 till January 2020
  Symptoms of posttraumatic stress disorder measured via screening tool (PTSD-7).

OTHER OUTCOMES:
Comorbidities | October 2019 till January 2020
  Relevant comorbidities (e.g. Diabetes, Hypertension, psychic comorbidities) will be taken from the medical record of the participants.
VAD Type | October 2019 till January 2020
  Information on implanted VAD type (HVAD, HMIII or other) will be taken from the medical record of the participants.
New York Heart Association (NYHA) classification | October 2019 till January 2020
  Information on New York Heart Association (NYHA) classification of the participants will be taken from their medical record.
VAD-related complications | October 2019 till January 2020
  Emerged VAD-related complications (e.g. neurologic events, major bleeding events, infections) will be taken from the patients' medical record.

CONTACTS AND LOCATIONS:
Overall Officials: Christiane Kugler, Prof. Dr., Study Director — University of Freiburg; Christiane Kugler, Prof. Dr., Principal Investigator — University of Freiburg
Locations (4):
- Germany (4):
  - University Heart Center Freiburg, Freiburg im Breisgau, Baden-Wurttemberg
  - Heart and Diabetes Center North Rhine-Westphalia, Bad Oeynhausen, North Rhine-Westphalia
  - Leipzig Heart Center, Leipzig, Saxony
  - German Heart Center, Berlin

REFERENCES:
- [Derived] Kugler C, Spielmann H, Albert W, Lauenroth V, Spitz-Koeberich C, Semmig-Koenze S, Staus P, Tigges-Limmer K; SELMA Study Group. Professional Employment in Patients on Ventricular Assist Device Support-A National Multicenter Survey Study. ASAIO J. 2024 May 1;70(5):348-355. doi: 10.1097/MAT.0000000000002124. Epub 2024 Jan 3. PMID 38170263
- [Derived] Spielmann H, Tigges-Limmer K, Albert W, Spitz-Koberich C, Semmig-Konze S, Staus P, Herrmann-Lingen C, Sandau KE, Okeson B, Geyer S, Kugler C; Selma Study Group. Health-Related Quality of Life in Patients With Ventricular Assist Device: Psychometric Evaluation of the German Version of the Quality of Life With a Ventricular Assist Device Questionnaire. J Cardiovasc Nurs. 2024 Nov-Dec 01;39(6):571-582. doi: 10.1097/JCN.0000000000001064. Epub 2023 Nov 22. PMID 37991265
- [Derived] Spielmann H, Albert W, Semmig-Konze S, Lauenroth V, Spitz-Koberich C, Staus P, Tigges-Limmer K, Kugler C; SELMA Study Group. High level of psychosocial adjustment in patients on ongoing ventricular assist device support in the years one to three after VAD implantation-A national multi-center Study. Heart Lung. 2024 Jan-Feb;63:92-97. doi: 10.1016/j.hrtlng.2023.10.003. Epub 2023 Oct 12. PMID 37837720
- [Derived] Kugler C, Spielmann H, Seemann M, Lauenroth V, Wacker R, Albert W, Spitz-Koeberich C, Semmig-Koenze S, von Cube M, Tigges-Limmer K. Self-management for patients on ventricular assist device support: a national, multicentre study: protocol for a 3-phase study. BMJ Open. 2021 May 5;11(5):e044374. doi: 10.1136/bmjopen-2020-044374. PMID 33952544
- [Derived] Spielmann H, Seemann M, Friedrich N, Tigges-Limmer K, Albert W, Semmig-Konze S, Spitz-Koberich C, Kugler C. Self-management with the therapeutic regimen in patients with ventricular assist device (VAD) support - a scoping review. Heart Lung. 2021 May-Jun;50(3):388-396. doi: 10.1016/j.hrtlng.2021.01.019. Epub 2021 Feb 20. PMID 33621837